CLINICAL TRIAL: NCT05032729
Title: Nutritional Intervention to Enhance Sleep Quality and Quantity in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-1911
Record Dates: First submitted 2021-08-13; First posted 2021-09-02 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Sleep; Physical Performance; Cognitive Performance; Balance
Keywords: nutrition; sleep; polysomnography; performance; exercise
MeSH Terms: conditions — Motor Activity | interventions — theanine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo beverage (Placebo Comparator): * Flavor
  * Non-nutritive sweetener
  * Color added to match whey appearance
  Interventions: Other: Placebo
- Higher tryptophan beverage (Experimental): * 2.7g high Glycemic Index Carbohydrate
  * 40g whey
  * 0.855g tryptophan
  * 660mg theanine
  * 53mcg 5'AMP
  * Non-nutritive sweetener
  * Flavor
  Interventions: Other: Trypophan, Theanine and 5'AMP
- Lower tryptophan beverage (Experimental): * 2.7g high Glycemic Index Carbohydrate
  * 30g whey
  * 0.641g tryptophan
  * 660mg theanine
  * 53mcg 5'AMP
  * Non-nutritive sweetener
  * Flavor
  Interventions: Other: Trypophan, Theanine and 5'AMP

INTERVENTIONS:
Other: Trypophan, Theanine and 5'AMP — 250 ml beverage consumed at 21:00 hours
  Arms: Higher tryptophan beverage; Lower tryptophan beverage
Other: Placebo — 250 ml beverage consumed at 21:00 hours, matched in appearance and taste to the active beverages
  Arms: Placebo beverage

SUMMARY:
The primary objective is to assess the impact of two nutritional interventions vs. placebo on objective and subjective sleep measures in athletes. Participants receive one beverage on each of three consecutive nights in a randomized manner. It is hypothesized the two nutritional interventions will result in significant improvements in sleep onset latency, and will not result in a negative impact on next-day cycling performance.

The secondary objective is to assess the impact of the nutritional interventions vs. placebo on next-morning performance (physical, cognitive function, and balance).

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-40 years old
* Healthy (assessed via the Exercise and Sports Science Australia (ESSA) survey
* Endurance trained (2 hours of training at least 3 days per week for a minimum of 3 years)
* Free from any known sleep disorders or disturbances as assessed by a Pittsburg Sleep Quality Index (PSQI score under 5)
* Must be willing to live/sleep at the Appleton Institute Sleep Laboratory for 4 (consecutive) nights/5 days (total 96 hours)
* Must be able to provide written informed consent upon having the study procedure explained to them verbally and in writing.
* Willing to be prohibited from consuming caffeine and alcohol during the entire stay at the sleep clinic and agree to eat only the standardized meals and snacks and drinks provided.

Exclusion Criteria:

* Subject has a clinically diagnosed sleeping disorder
* Subject has a change in medication over the duration of the study that is known to affect sleep
* Subject has a current illness that would affect sleep
* Subject has a current injury that would prevent him from giving maximal effort during the next-morning performance task
* Participation in another clinical trial within the past 30 days or another PepsiCo/GSSI study within the past 6 months

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological males due to the influence that menstrual cycle may have on sleep and the study aims to investigate previous findings involving male only participants
Enrollment: 19 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Total Sleep Time (TST) | Time from sleep onset to 8:00 a.m.
  Measured in minutes during polysomnography. Longer is better.
Wake After Sleep Onset (WASO) | From sleep onset till 8:00 a.m.
  Occurrences measured in minutes during polysomnography. None or less are better.
Sleep Efficiency (SE) | From sleep onset to 8:00 a.m.
  Measured as a % of time asleep over time in bed during polysomnography. Higher efficiency is better
Sleep Onset Latency (SOL) | Transition from wakefulness to sleep
  Measured in minutes during polysomnography. Shorter time to onset is better.
Rapid Eye Movement (REM) Latency | From sleep onset to REM sleep
  Measured in minutes during polysomnography. Shorter time to REM is better.
Sleep stage 3 Latency | From sleep onset to deep sleep
  Measured in minutes during polysomnography. Shorter time to stage 3 deep sleep is better.
Sleep stage 1, 2, 3 AND REM | Measured continuously throughout the night from sleep onset to 8 a.m.
  Measured in minutes during polysomnography. Normal stage pattern is better.
Arousals | From sleep onset to 8 a.m.
  Measured as a count during polysomnography. Less arousals are better.
Awakenings | From sleep onset to 8 a.m.
  Measured as a count during polysomnography. Less awakenings are better.
Stage shifts | From sleep onset to 8 a.m.
  Measured as a count during polysomnography. Normal amount of stage shifts are better.
Subjective Karolinska Sleepiness Scale (KSS) | Every thirty minutes from 20:00 p.m. until 22:30 p.m.
  Subjective arousal level at present state rated 1 (extremely alert) to 9 (Very sleepy, great effort to keep awake). Sleepiness before bed is better.
(Subjective) Perceived Sleep Quality | 08:30 a.m. following polysomnography
  Rated from 1 (very good) to 5 (poor). Lower number is better.
(Subjective) Sleep Quantity | 08:30 a.m. following polysomnography
  Measured in hours and minutes. Higher number is better.
(Subjective) Sleep Onset Latency | 08:30 a.m. following polysomnography
  Measured in hours and minutes. Lower number is better.

SECONDARY OUTCOMES:
Exercise performance: power output | During a 10 minute time trial cycling exercise performance testing at 9:30 a.m.
  Cycle ergometer to measure power output in watts, with instructions to give maximal effort. Higher watts are better.
Exercise performance: perceived exertion | During a 10 minute time trial cycling exercise performance testing at 9:30 a.m.
  Rating of perceived exertion (RPE) on a scale of 6 (lower) to 20 (higher) intensity levels.
Exercise performance: heart rate | During a 10 minute time trial cycling exercise performance testing at 9:30 a.m.
  Measured in beats per minute (bpm) by heart rate monitor
Cognitive performance: sustained attention | 10 minute testing period at 9 a.m. Higher performance is better.
  Psychomotor vigilance reaction time task (PVT-192) handheld ambulatory monitoring
Subjective alertness | 9 a.m. before cognitive performance attention testing.
  Rated on visual analog scale from 0 (feeling not at all alert) to 100 (feeling completely alert). Feeling more alert is better.
Subjective self-perceived capacity to be fast on cognitive test | 9 a.m. before cognitive performance attention testing
  Rated on visual analog scale from 0 (expecting to not respond fast at all) to 100 (expecting to respond very fast). Better or worse not applicable.
Subjective self-perceived capacity to be accurate on cognitive test | 9 a.m. before cognitive performance attention testing
  Rated on visual analog scale from 0 (expecting to not respond accurately at all) to 100 (expecting to respond very accurately). Better or worse not applicable.
Balance | 9 a.m. before cognitive performance attention testing.
  Postural sway area 95cm/2 measured by computerized force platform. Less sway is better.

CONTACTS AND LOCATIONS:
Overall Officials: Shona Halson, PhD, Principal Investigator — Appleton Institute CQUniversity, School of Medical, Health, and Applied Sciences, Adelaide Campus and Australian Catholic University
Locations (1):
- Appleton Institute CQUniversity, School of Medical, Health, and Applied Sciences, Adelaide Campus, Wayville, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No